CLINICAL TRIAL: NCT07305363
Title: The SELIC Trial Seladelpar for the Treatment of Ischemic Cholangiopathy: An Open-Label, Single-Arm, Investigator-Initiated Study
Brief Title: A Prospective, Open-label, Single-arm, Investigator-initiated Study (SELIC) to Evaluate the Efficacy and Safety of Seladelpar in Adult Liver Transplant Recipients With Ischemic Cholangiopathy (IC).
Acronym: SELIC
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Veeral Ajmera, Associate Professor Of Clinical, Medicine, University of California, San Diego
Other Study IDs: Clinical Protocol #:NRC-2023-1
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant; Complications; Ischemic Cholangiopathy
MeSH Terms: interventions — seladelpar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Seladelpar: Seladelpar 10 mg orally once daily for 52 weeks
  Interventions: Drug: Seladelpar

INTERVENTIONS:
Drug: Seladelpar — Seladelpar is a selective peroxisome proliferator-activated receptor delta (PPAR-δ) agonist

SUMMARY:
A prospective, open-label, single-arm, investigator-initiated study (SELIC) to evaluate the efficacy and safety of seladelpar in adult liver transplant recipients with Ischemic cholangiopathy (IC).

DETAILED DESCRIPTION:
Ischemic cholangiopathy (IC) is a serious complication after liver transplantation, particularly in recipients of donation after circulatory death grafts, and is associated with cholestasis, biliary strictures, and graft dysfunction. No approved pharmacologic therapies currently exist. Seladelpar, a selective peroxisome proliferator-activated receptor delta (PPAR-δ) agonist recently approved for primary biliary cholangitis, reduces bile acid synthesis and inflammation and has demonstrated antifibrotic activity, making it a promising candidate for IC. We designed a prospective, open-label, single-arm, investigator-initiated study (SELIC) to evaluate the efficacy and safety of seladelpar in adult liver transplant recipients with IC. Ten patients will receive seladelpar 10 mg orally once daily for 52 weeks. Outcomes will be compared to historical controls identified from the same institution. The primary endpoint is percent change in serum alkaline phosphatase (ALP) from baseline to Week 26. Additional outcomes include ERCP utilization, liver allograft loss, and safety assessed by adverse event and laboratory monitoring and drug discontinuation rates. This pilot study will provide the first prospective data on seladelpar in IC and may establish preliminary evidence for a novel therapeutic approach to reduce cholestasis, improve symptoms, and preserve graft function in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age ≥ 18 and < 80 years
2. Diagnosis of ischemic cholangiopathy defined as non-anastomotic biliary strictures confirmed by imaging (ERCP, MRI, percutaneous cholangiogram)
3. Cholestasis noted by elevated alkaline phosphatase (ALP) and gamma glutamyl transferase (GGT)
4. Imaging and clinical findings present at least 4 weeks after but within 12 months of liver transplantation
5. No recent hospitalization within 2 weeks before enrollment to ensure clinical stability

Exclusion Criteria:

1. Decompensated liver disease, including but not limited to ascites requiring paracentesis, hepatic encephalopathy, or variceal bleeding.
2. Pregnancy or breastfeeding.
3. Current or recent (within 30 days) use of other investigational agents or fenofibrate.
4. Current or recent (within 30 days) use of cyclosporine
5. Known hypersensitivity or contraindication to seladelpar or its excipients.
6. Severe concomitant illness (renal, cardiac, or other systemic condition) that, in the investigator's judgment, would interfere with study participation or interpretation of results.
7. ALT > 150 IU/L.
8. AST > 150 IU/L.
9. Total bilirubin > 5 mg/dL at screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet study eligibility criteria will be recruited from UCSD's liver transplant clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
serum alkaline phosphatase (ALP) | 26 weeks
  Determine the effect of seladelpar on serum alkaline phosphatase (ALP) from baseline to week 26

IPD SHARING:
Plan to Share IPD: Undecided